CLINICAL TRIAL: NCT06031987
Title: Long-term Effects of Flash Glucose Monitoring System in Patients With Gestational Diabetes
Acronym: GDMLIBRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Cheol-Young Park, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GDMLIBRE
Record Dates: First submitted 2022-10-21; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Intervention Model Description: randomized, parallel, open labeled study
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SMBG arm (Active Comparator): Self Monitoring of Blood Glucose group
  Interventions: Device: CareSens N (iSENS)
- CGMS arm (Experimental): Continuous glucose monitoring system, CGM
  Interventions: Device: Freestyle Libre (Abbott)

INTERVENTIONS:
Device: CareSens N (iSENS) — Control group is asked to perform SMBG (4 times or more per day).
  Arms: SMBG arm
Device: Freestyle Libre (Abbott) — CGM group is asked to scan CGM (4 times or more per day).
  Arms: CGMS arm

SUMMARY:
The purpose of this study is to report the glycemic control effect and clinical safety and effectiveness of mother and fetus when using a continuous glucose monitoring system (CGM) [Freestyle Libre] for a long period of time compared to self monitoring blood glucose(SMBG) in gestational diabetes patients.

DETAILED DESCRIPTION:
The investigators plan to conduct a randomized clinical trial among patients with Gestational Diabetes Mellitus (GDM). The intervention group will use Continuous Glucose Monitoring (CGM) throughout the study period, scanning four or more times per day. The control group will be instructed to perform Self-Monitoring Blood Glucose (SMBG), also four or more times per day.

Eligible participants are those within 24 to 30 weeks of gestation (Visit 0). These subjects will undergo a 1-week run-in period, during which they will wear a retrospective CGM device and perform SMBG four or more times daily as a part of the screening process (Visit 1).

Following the run-in period, subjects will be randomly assigned to either the CGM group (using the Freestyle Libre device) or the Control group (using SMBG). Members of the control group will be asked to perform SMBG four or more times daily, while those in the CGM group will be instructed to scan their CGM four or more times per day.

Participants will have clinic visits at intervals ranging from 2 to 4 weeks, the frequency of which will be determined at the discretion of the attending physician (Visits 2, 2', 2'', 2''', 2''').

Upon reaching gestational age 34-35 weeks (Visit 3), members of the control group will begin to wear a retrospective CGM device until they reach gestational age 36 weeks (Visit 4).

After 6-12 weeks from delivery, subjects will be asked to visit the clinic again and undergo a 75g Oral Glucose Tolerance Test (OGTT) (Visit 5).

For the purposes of data analysis and outcome determination, the most recent 1-week CGM data collected at Visit 4 will be used for both groups.

ELIGIBILITY:
[Inclusion Criteria]

1. 19-40 aged female
2. Gestational diabetes diagnosed at 24 to 28 weeks of pregnancy screening (stage 1 or stage 2 approach)

   * 2-1.Screening one-step approach (75g oral glucose tolerance test, diagnosed when one or more of the following)

     * Fasting blood glucose 92 mg/dL or higher
     * Blood glucose 180 mg/dL or higher 1 hour after glucose loading
     * Blood glucose of 153 mg/dL or higher 2 hours after glucose loading
   * 2-2. Screening two-step approach (50 g oral glucose tolerance test then,100g oral glucose tolerance test)

     * If the blood glucose level is 140 mg/dL or higher for 1 hour after the 50g oral glucose tolerance test,
     * 100g oral glucose tolerance test 2 or more of the following

       1. Fasting blood glucose 95mg/dL or higher
       2. Blood glucose 180mg/dL or higher 1 hour after glucose loading
       3. Blood glucose of 155 mg/dL or higher 2 hours after glucose loading
       4. Blood glucose of 140 mg/dL or higher 3 hours after glucose loading
3. Singleton Pregnancy

[Exclusion Criteria]

- pregestational diabetes (Overt diabetes)

1. Diabetes Before Pregnancy
2. At least one of the following at the first prenatal visit

   * Fasting blood glucose 126mg/dL or higher
   * Random blood glucose 200mg/dL or higher

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gestational Diabetes
Enrollment: 100 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-01-26 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
63-140 mg/dL Time in Range | at visit 4(gestational age 36weeks)
  63-140 mg/dL Time in Range evaluated for 1 week before Visit4 visit

SECONDARY OUTCOMES:
AbA1C (%) | at visit 4(gestational age 36weeks)
  HbA1C evaluated at visit 4
Glycated Albumin(g/dL) | at visit 4(gestational age 36weeks)
  Glycated Albumin evaluated at visit 4
>180 mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  >180 mg/dL Time in Range evaluated for 1 week before Visit4
>140 mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  >140 mg/dL Time in Range evaluated for 1 week before Visit4
>120 mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  >120 mg/dL Time in Range evaluated for 1 week before Visit4
<63mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  <63mg/dL Time in Range evaluated for 1 week before Visit4
<54mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  <54mg/dL Time in Range evaluated for 1 week before Visit4
63-120mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  63-120mg/dL Time in Range evaluated for 1 week before Visit4
Night time Blood glucose (0AM-6AM) 63-94 mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  Night time Blood glucose (0AM-6AM) 63-94 mg/dL Time in Range evaluated for 1 week before Visit4
Night time Blood glucose (0AM-6AM) ≥95 mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  Night time Blood glucose (0AM-6AM) ≥95 mg/dL Time in Range evaluated for 1 week before Visit4
Night time Blood glucose (0AM-6AM) <63 mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  Night time Blood glucose (0AM-6AM) <63 mg/dL Time in Range evaluated for 1 week before Visit4
Night time Blood glucose (0AM-6AM) <54 mg/dL Time in Range | 1 week before Visit4 (gestational age 36weeks)
  Night time Blood glucose (0AM-6AM) <54 mg/dL Time in Range evaluated for 1 week before Visit4
Overall average blood glucose level | 1 week before Visit4 (gestational age 36weeks)
  Overall average blood glucose level evaluated for 1week before visit4
Overall average Night time Blood glucose (0AM-6AM) level | 1 week before Visit4 (gestational age 36weeks)
  Overall average Night time Blood glucose (0AM-6AM) level evaluated for 1week before visit4
Overall average During the day time blood glucose (6AM-12PM) level | 1 week before Visit4 (gestational age 36weeks)
  Overall average During the day time blood glucose (6AM-12PM) level evaluated for 1week before visit4
Frequency of severe hypoglycemia(Hypoglycemia requiring help from others) | From visit 1 to visit 4(Gestational age 25-31 weeks to Gestational age 36 week)
  Frequency of severe hypoglycemia during the study period hyperglycemia requiring help from others)
glucose variability | 1 week before Visit4(gestational age 36weeks)
  glucose variability evaluated for 1week before visit4 (MAGE,SD,CV)
rate of insulin treatment | From visit 1 to visit 4 (Gestational age 25-31 weeks to Gestational age 36 week)
  rate of insulin treatment
Estimation A1c of continuous blood glucose measurement for 1 week before Visit4 visit | 1 week before Visit4(Gestational age 36 week)
  Estimation A1c of continuous blood glucose measurement for 1 week before Visit4 visit
Total daily insulin requirements (evaluated at every visit) | From visit 1 to visit 4(Gestational age 25-31 weeks to Gestational age 36 week)
  Total daily insulin requirements (evaluated at every visit)
Satisfaction Questionnaire | Visit 1 (Gestational age 25-31 weeks) , Visit 4 (Gestational age 36 week)
  Satisfaction Questionnaire(DTSQ) ,Score: min0 ~max 48, higher scores mean a better outcome
C-section rate | during the study period (Gestational age 25-31 weeks to Pospartum 6-12 weeks)
  C-section rate
preeclampsia rate | during the study period (Gestational age 25-31 weeks to Pospartum 6-12 weeks)
  preeclampsia rate
preeclampsia or gestational hypertension rate | during the study period (Gestational age 25-31 weeks to Pospartum 6-12 weeks)
  preeclampsia or gestational hypertension rate
the rate of preterm birth | during the study period (Gestational age 25-31 weeks to Pospartum 6-12 weeks)
  the rate of preterm birth
Weight gain during the study period | during the study period (Gestational age 25-31 weeks to Pospartum 6-12 weeks)
  Weight gain during the study period
Average daily blood glucose measurements during the study period | during the study period (Gestational age 25-31 weeks to Pospartum 6-12 weeks)
  Freestyle Libre scans, SMBG
Changes in Microbiome | during the study period (Gestational age 25-31 weeks to Pospartum 6-12 weeks)
  Changes in Microbiome
Rate of transition to type 2 diabetes | at post partum (6-12 weeks after delivery)
  Rate of transition to type 2 diabetes
Rate of transition to Glucose intolerance (prediabetes and/or diabetes) | at post partum (6-12 weeks after delivery)
  Rate of transition to Glucose intolerance (prediabetes and/or diabetes)
Rate of transition to Impaired fasting glucose (IFG) and/or diabetes | at post partum (6-12 weeks after delivery)
  Rate of transition to Impaired fasting glucose (IFG) and/or diabetes
Rate of transition to Impaired fasting glucose (IGT) and/or diabetes | at post partum (6-12 weeks after delivery)
  Rate of transition to Impaired fasting glucose (IGT) and/or diabetes
75g OGTT hourly blood glucose | at post partum (6-12 weeks after delivery)
  75g OGTT hourly blood glucose
hemoglobinA1C | at post partum (6-12 weeks after delivery)
  hemoglobinA1C
glycated albumin | at post partum (6-12 weeks after delivery)
  glycated albumin
Insulin resistance index (HOMA-IR) | at post partum (6-12 weeks after delivery)
  HOMA-IR (no unit, higher score means a worse outcome)
Insulin resistance index (Matsuda index) | at post partum (6-12 weeks after delivery)
  Matsuda index (no unit, higher score means a better outcome)
Insulin secretion ability index (HOMA-beta) | at post partum (6-12 weeks after delivery)
  HOMA-beta(no unit, higher score means a better outcome)
Insulin secretion ability index (Insulinogenic index) | at post partum (6-12 weeks after delivery)
  Insulinogenic index(no unit, higher score means a better outcome)
Insulin Composite index(Oral disposition index) | at post partum (6-12 weeks after delivery)
  Oral disposition index(no unit, higher score means a better outcome)
Insulin Composite index(disposition index) | at post partum (6-12 weeks after delivery)
  disposition index(no unit, higher score means a better outcome)
weight change | at post partum (6-12 weeks after delivery)
  weight change
Change in Bioelectric impedance analysis (BIA) | at post partum (6-12 weeks after delivery)
  Change in Bioelectric impedance analysis (BIA)
fetal: childbirth weight | at Delivery
  fetal: childbirth weight
fetal: Macrosomia ( > 4000 g) | at Delivery
  fetal: Macrosomia ( > 4000 g)
fetal:Large for gestational age ( > 90th percentile for age) | at Delivery
  fetal:Large for gestational age ( > 90th percentile for age)
fetal:Small for gestational age ( < 10th percentile for age) | at Delivery
  fetal:Small for gestational age ( < 10th percentile for age)
fetal:Neonatal glucose level | at Delivery
  fetal:Neonatal glucose level
fetal:NICU admission | at Delivery
  fetal:NICU admission
fetal:birth trauma (including shoulderdystocia, clavicle fracture or Erb's palsy) | at Delivery
  fetal:birth trauma (including shoulderdystocia, clavicle fracture or Erb's palsy)
fetal:Pre-term birth | at Delivery
  fetal:Pre-term birth
fetal:Apgar score | at Delivery
  score: min 0 ~ max 10, higher scores mean a better outcome
fetal:Meconium aspiration | at Delivery
  fetal:Meconium aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Cheol-Young Park, MD, Principal Investigator — KangbukSamsung Hospital
Locations (1):
- Kangbuk Samsung hospital, Seoul, South Korea

REFERENCES:
- [Result] Cespedes EM, Hu FB, Tinker L, Rosner B, Redline S, Garcia L, Hingle M, Van Horn L, Howard BV, Levitan EB, Li W, Manson JE, Phillips LS, Rhee JJ, Waring ME, Neuhouser ML. Multiple Healthful Dietary Patterns and Type 2 Diabetes in the Women's Health Initiative. Am J Epidemiol. 2016 Apr 1;183(7):622-33. doi: 10.1093/aje/kwv241. Epub 2016 Mar 2. PMID 26940115
- [Result] Guariguata L, Linnenkamp U, Beagley J, Whiting DR, Cho NH. Global estimates of the prevalence of hyperglycaemia in pregnancy. Diabetes Res Clin Pract. 2014 Feb;103(2):176-85. doi: 10.1016/j.diabres.2013.11.003. Epub 2013 Dec 1. PMID 24300020
- [Result] Kim KS. The importance of treating mild hyperglycemia in pregnant women with diabetes. Korean J Intern Med. 2018 Nov;33(6):1079-1080. doi: 10.3904/kjim.2018.351. Epub 2018 Oct 30. No abstract available. PMID 30396252
- [Result] Koo BK, Lee JH, Kim J, Jang EJ, Lee CH. Prevalence of Gestational Diabetes Mellitus in Korea: A National Health Insurance Database Study. PLoS One. 2016 Apr 5;11(4):e0153107. doi: 10.1371/journal.pone.0153107. eCollection 2016. PMID 27046149
- [Result] DeSisto CL, Kim SY, Sharma AJ. Prevalence estimates of gestational diabetes mellitus in the United States, Pregnancy Risk Assessment Monitoring System (PRAMS), 2007-2010. Prev Chronic Dis. 2014 Jun 19;11:E104. doi: 10.5888/pcd11.130415. PMID 24945238
- [Result] McIntyre HD, Catalano P, Zhang C, Desoye G, Mathiesen ER, Damm P. Gestational diabetes mellitus. Nat Rev Dis Primers. 2019 Jul 11;5(1):47. doi: 10.1038/s41572-019-0098-8. PMID 31296866
- See also: Hasain Z, Mokhtar NM , Kamaruddin NA, Mohamed Ismail NA, Razalli NH, Gnanou JV, et al. Gut Microbiota and Gestational Diabetes Mellitus: A Review of Host Gut Microbiota Interactions and Their Therapeutic Potential. Front Cell Infect Microbiol [Internet]. — https://www.frontiersin.org/articles/10.3389/fcimb.2020.00188/full